CLINICAL TRIAL: NCT00136279
Title: RCT of Tobacco Use Prevention and Sexual Risk Reduction Interventions for Parents of African American and Latino Youth in Middle School
Brief Title: Linking Lives: Building Quality Parent Components for School-Based Health Programs in Middle Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Columbia University (Other)
Responsible Party: Vincent Guilamo-Ramos, Columbia University School of Social Work
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CDC-NCCDPHP-3486; U87/CCU220155-05
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-01

CONDITIONS: Smoking; Sexual Behavior
Keywords: adolescent behavior; sexual behavior; smoking; parents; communication; health education; schools; Sexual initiation
MeSH Terms: conditions — Smoking; Sexual Behavior; Adolescent Behavior; Communication; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- School plus parent (Experimental): Adolescents receive school-based curriculum (either Project TNT or Making a Difference) and mothers receive the Linking Lives curriculum
  Interventions: Behavioral: Linking Lives parent-based intervention
- School-only (Active Comparator): Adolescents receive school-based curriculum and parents received a control curriculum on helping their child choose a high school
  Interventions: Behavioral: Linking Lives parent-based intervention
- Parent-Only (Experimental): In the sex risk reduction portion of the study only, a second experimental group consisted of parents receiving the Linking Lives intervention and adolescents receiving no in-school intervention
  Interventions: Behavioral: Linking Lives parent-based intervention

INTERVENTIONS:
Behavioral: Linking Lives parent-based intervention — Parent intervention consists of mothers attending two, 2.5 hour-long, face-to-face sessions at the school during which they are given an intervention manual, two homework assignments, and a manual for their adolescent. Parents also receive two booster telephone calls approximately one-month and six-months after completing the intervention. As part of the comparison condition, school-based interventions for adolescents also consist of two, 2.5 hour-long, face-to-face sessions at schools during which they complete either the Project TNT intervention for preventing tobacco use or the Making a Difference intervention for reducing sexual risk behavior.

SUMMARY:
The purpose of this study is to develop and evaluate the effectiveness of a parent-based intervention that can be implemented in conjunction with existing school-based programs designed to prevent or reduce sexual risk behavior or to prevent or reduce tobacco use in young adolescents. The parent programs are expected to have effects on adolescent behavior over and above the effects of the school-based programs.

DETAILED DESCRIPTION:
Although parent-based programs have shown promise in reducing adolescent risk behavior, few have been rigorously evaluated and shown to be effective. Recruitment and retention of parents into lengthy workshops has been a problem and few programs have been developed specifically for inner-city, minority populations who are at greatest risk for a number of adverse health outcomes. Linking Lives was designed to address these issues.

Parent Intervention. The primary feature of the parent component is a written manual distributed in modules to mothers that teaches them how to communicate effectively with their children about sex or tobacco risk behaviors and how to improve their relationships with their children. This is accompanied by two face-to-face intervention sessions for mothers, during which they are given the intervention materials and an opportunity to participate in role playing activities with other parents, and by regular contact by trained parent volunteers to determine if the parent has implemented the manual contents. Mothers and their adolescents attend Linking Lives events together at the school in the evenings and on weekends during which time adolescents attend their own intervention sessions at the same time mothers are attending theirs (mothers in the control condition participate in sessions on helping their children choose a high school).

Sample. Nine middle schools in the Bronx, New York and two schools in the Harlem neighborhood of New York are participating in the study. The schools are located in communities that are financially disadvantaged. Approximately 70% of the students in the schools are Latino and 30% are African American. A total of 4,750 adolescents and their mothers will participate in the study, 1,900 for tobacco and 2,850 for sexual risk reduction. Students are randomly sampled and their parent is contacted regarding family participation in the study.

Evaluation. Based on input from elicitation studies, focus groups with adolescents and mothers, a pre-intervention survey of 668 mother-adolescent pairs, a psychometric study for both English- and Spanish-language instruments, feedback from community and school leaders, and a scientific panel of experts, the instruments, manuals and intervention protocol have been developed. All measures and intervention materials have been developed in English and in Spanish. The evaluation includes a baseline, 3-month post-test and a 15-month delayed post-test assessment of adolescents and mothers. For tobacco, within schools, students will be randomly assigned to an experimental group (school-based curriculum plus parent component) or a control group (school-based curriculum only). For sexual risk reduction, students will be randomly assigned to the combined experimental condition (school-based curriculum plus parent component), a parent-only experimental condition (parent component is distributed to mothers, but no school component is delivered) or a control group (school-based curriculum only).

ELIGIBILITY:
Inclusion Criteria:

* African American or Latino
* 6th or 7th grade students
* Residential mothers or primary female caregivers

Exclusion Criteria:

* 8th grade students
* Fathers or primary male caregivers

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9510 (Estimated)
Dates: Start 2004-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Self-reported ever had sex or ever smoked a cigarette | 3-month and 15-month follow-up

SECONDARY OUTCOMES:
Intentions to have sex or to smoke cigarettes | 3-month and 15-month follow-up
Age at first intercourse or first cigarette | 3-month and 15-month follow-up
Condom use at last sex | 3-month and 15-month follow-up
Contraceptive use at last sex | 3-month and 15-month follow-up
Maternal monitoring and supervision | 3-month and 15-month follow-up
Maternal Communication about smoking cigarettes or sexual intercourse | 3-month and 15-month follow-up
Quality of maternal communication | 3-month and 15-month follow-up
Self-reported regular cigarette smoking | 3-month and 15-month follow-up
Intentions to smoke marijuana | 3-month and 15-month follow-up
Ever smoked marijuana | 3-month and 15-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Guilamo-Ramos, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University School of Social Work, New York, New York, United States